CLINICAL TRIAL: NCT02879110
Title: A 12-weeks, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy, Safety and Related Mechanism of Sulforaphane in Treatment of Autism Spectrum Disorder
Brief Title: A 12-weeks Study to Evaluate Sulforaphane in Treatment of Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Collaborators: Davis family funding (Unknown); University of California (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Jian-Jun Ou, Assistant researcher, Central South University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASD201512
Record Dates: First submitted 2016-08-15; First posted 2016-08-25 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Autism Spectrum Disorder
Keywords: Sulforaphane; clinic trial; Autism Spectrum Disorder; Efficacy; Safety; Mechanism
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — sulforaphane; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sulforaphane group (Experimental): The patients will take sulforaphane for 12 weeks.
  Interventions: Dietary Supplement: Sulforaphane
- Placebo group (Placebo Comparator): The patients will take placebo for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Sulforaphane — Sulforaphane (SFN) is a compound within the isothiocyanate group of organosulfur compounds. It is obtained from cruciferous vegetables such as broccoli, Brussels sprouts or cabbages.
  Other Names: 85313323
  Arms: Sulforaphane group
Other: Placebo — Placebo tablet is composed of starch.
  Other Names: Starch tablet
  Arms: Placebo group

SUMMARY:
In this proposed study, the investigators will evaluate the the efficacy, safety and related mechanism of sulforaphane in treatment of autism spectrum disorder (ASD). The study will recruit 120 ASD patients, then these patients will be randomized to sulforaphane group or placebo group (60 patients per arm) for 12 weeks clinic trial. Clinical efficacy and safety assessment will be done at screen/baseline, 4 week, 8 week and 12 week. The specific aims are to compare sulforaphane versus placebo on: 1) clinical core symptoms; 2) other behavioral problems and adaptive behaviors. Biological samples also will be collected, and stored to research related mechanisms.

DETAILED DESCRIPTION:
In this proposed study, the investigators will evaluate the the efficacy, safety and related mechanism of sulforaphane in treatment of autism spectrum disorder (ASD). The study will recruit 120 ASD patients, then these patients will be randomized to sulforaphane group or placebo group (60 patients per arm) for 12 weeks clinic trial. Clinical efficacy and safety assessment will be done at screen/baseline, 4 week, 8 week and 12 week. The specific aims are to compare sulforaphane versus placebo on: 1) clinical core symptoms; 2) other behavioral problems and adaptive behaviors. The investigators hypothesize that (1) sulforaphane is superior to placebo in the treatment of clinical symptoms in patients with ASD, measured by the Social Responsiveness Scale, Aberrant Behavior Checklist, Repetitive Behavior Scale - Revised and Ohio State University Autism Clinical Global Impression; (2) sulforaphane is superior to placebo in the treatment of other behavioral problems and adaptive behaviors patients with ASD, measured by Achenbach's Child Behavior Checklist and Adaptive Behavior Assessment System, Second Edition; and (3) Biological samples will be collected, and stored so that the hypothesis sulforaphane may alter oxidative stress indexes or inflammatory biomarkers, and influence histone deacetylase inhibitor mechanism or inflammatory mechanism et al that may be significantly correlated with clinical improvement.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 3 to 15 years.
2. Meet DSM-V diagnostic criteria for autism spectrum disorder, and been checked with Autism Diagnostic Interview-Revised (ADI-R) and Autism Diagnostic Observation Schedule (ADOS).

Exclusion Criteria:

1. With severe physical disease (i.e. congenital heart disease, thyroid disease, diseases with severe abnormality of liver or kidney function, diseases with abnormality vision or hearing et al.)
2. With severe central nervous system disease (i.e. epilepsy et al).
3. With other specific genetic syndromes (i.e. Fragile-X syndrome, Down's syndrome et al.)

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2016-08; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
The change of social impairments of children with autism spectrum disorder | At baseline, 4 week, 8 week and 12 week/endpoint
  Social impairments are measured by Social Responsiveness Scale

SECONDARY OUTCOMES:
The change of rigid interests and behaviors of children with autism spectrum disorder | At baseline, 4 week, 8 week and 12 week/endpoint
  Rigid interests and behaviors are measured by Repetitive Behavior Scale - Revised
The change of clinical symptoms of children with autism spectrum | At baseline, 4 week, 8 week and 12 week/endpoint
  Clinical symptoms are measured by Aberrant Behavior Checklist
The change of other behavioral problems of children with autism spectrum | At baseline, 4 week, 8 week and 12 week/endpoint
  Other behavioral problems are measured by Achenbach's Child Behavior Checklist
The change of adaptive behaviors of children with autism spectrum | At baseline, 4 week, 8 week and 12 week/endpoint
  Adaptive behaviors are measured by Adaptive Behavior Assessment System, Second Edition
The change of clinical general impression of children with autism spectrum | At baseline, 4 week, 8 week and 12 week/endpoint
  Clinical general impression is measured by Ohio State University Autism Clinical Global Impression
The change of heart rate as measured by stopwatch | At baseline and 12 week/endpoint
The change of weight as measured by weighing-machine | At baseline and 12 week/endpoint
The change of height as measured by Height measurement tools | At baseline and 12 week/endpoint
The change of blood routine test as tested by clinical laboratory | At baseline and 12 week/endpoint
The change of fasting blood-glucose as tested by clinical laboratory | At baseline and 12 week/endpoint
The change of blood lipid as tested by clinical laboratory | At baseline and 12 week/endpoint
The change of liver function as tested by clinical laboratory | At baseline and 12 week/endpoint
The change of kidney function as tested by clinical laboratory | At baseline and 12 week/endpoint
The change of thyroid function as tested by clinical laboratory | At baseline and 12 week/endpoint
The change of HBV test as tested by clinical laboratory | At baseline and 12 week/endpoint
The change of helicobacter pylori test as tested by clinical laboratory | At baseline and 12 week/endpoint
The change of urine routine test as tested by clinical laboratory | At baseline and 12 week/endpoint
Number of participants with treatment-related adverse events as assessed by Systematic Assessment for Treatment Emergent Effects | At 4 week, 8 week and 12 week/endpoint

OTHER OUTCOMES:
The change of Oxidative stress indexes as tested by Oxidative stress indexes detection kit | At baseline and 12 week/endpoint
The change of Epigenetics indicators as tested by Epigenetics indicators | At baseline and 12 week/endpoint
The change of Cytokines & Chemokines as tested by Cytokines & Chemokines detection kit | At baseline and 12 week/endpoint
The change of Metabolites as tested by Metabolites detection kit | At baseline and 12 week/endpoint
The change of RNA expression as tested by RNA expression detection kit | At baseline and 12 week/endpoint
The change of intestinal microflora as tested by Metagenomic technique | At baseline and 12 week/endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Jingping Zhao, M.D., Ph. D., Study Chair — Central South University; Jianjun Ou, M.D., Ph. D., Study Director — Central South University; Hua Jin, M.D., Ph. D., Study Director — Department of Psychiatry, University of California; Fengyu Zhang, Ph.D., Principal Investigator — Global Clinical and Translational Research Institute; Daomeng Cheng, M.D., Principal Investigator — Guangzhou Huiai Hospital; Renrong Wu, M.D.,Ph.D, Principal Investigator — Central South University; John M Davis, M.D.,Ph.D, Study Director — Department of Psychiatry, University of Illinoisat at Chicago
Locations (2):
- China (2):
  - Guangzhou Huiai Hospital, Guangzhou, Guangdong
  - The second Xiangya hospital of central south university, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Foley AG, Cassidy AW, Regan CM. Pentyl-4-yn-VPA, a histone deacetylase inhibitor, ameliorates deficits in social behavior and cognition in a rodent model of autism spectrum disorders. Eur J Pharmacol. 2014 Mar 15;727:80-6. doi: 10.1016/j.ejphar.2014.01.050. Epub 2014 Jan 31. PMID 24486700
- [Background] Houghton CA, Fassett RG, Coombes JS. Sulforaphane: translational research from laboratory bench to clinic. Nutr Rev. 2013 Nov;71(11):709-26. doi: 10.1111/nure.12060. Epub 2013 Oct 22. PMID 24147970
- [Background] Moldrich RX, Leanage G, She D, Dolan-Evans E, Nelson M, Reza N, Reutens DC. Inhibition of histone deacetylase in utero causes sociability deficits in postnatal mice. Behav Brain Res. 2013 Nov 15;257:253-64. doi: 10.1016/j.bbr.2013.09.049. Epub 2013 Oct 5. PMID 24103642
- [Background] Foley AG, Gannon S, Rombach-Mullan N, Prendergast A, Barry C, Cassidy AW, Regan CM. Class I histone deacetylase inhibition ameliorates social cognition and cell adhesion molecule plasticity deficits in a rodent model of autism spectrum disorder. Neuropharmacology. 2012 Sep;63(4):750-60. doi: 10.1016/j.neuropharm.2012.05.042. Epub 2012 Jun 6. PMID 22683514
- [Background] Montes G, Halterman JS. Association of childhood autism spectrum disorders and loss of family income. Pediatrics. 2008 Apr;121(4):e821-6. doi: 10.1542/peds.2007-1594. PMID 18381511
- [Background] Montes G, Halterman JS. Child care problems and employment among families with preschool-aged children with autism in the United States. Pediatrics. 2008 Jul;122(1):e202-8. doi: 10.1542/peds.2007-3037. PMID 18595965
- [Background] Mugno D, Ruta L, D'Arrigo VG, Mazzone L. Impairment of quality of life in parents of children and adolescents with pervasive developmental disorder. Health Qual Life Outcomes. 2007 Apr 27;5:22. doi: 10.1186/1477-7525-5-22. PMID 17466072
- [Background] Myzak MC, Tong P, Dashwood WM, Dashwood RH, Ho E. Sulforaphane retards the growth of human PC-3 xenografts and inhibits HDAC activity in human subjects. Exp Biol Med (Maywood). 2007 Feb;232(2):227-34. PMID 17259330
- [Background] Ou JJ, Shi LJ, Xun GL, Chen C, Wu RR, Luo XR, Zhang FY, Zhao JP. Employment and financial burden of families with preschool children diagnosed with autism spectrum disorders in urban China: results from a descriptive study. BMC Psychiatry. 2015 Jan 22;15:3. doi: 10.1186/s12888-015-0382-4. PMID 25608486
- [Background] Rossignol DA, Frye RE. A review of research trends in physiological abnormalities in autism spectrum disorders: immune dysregulation, inflammation, oxidative stress, mitochondrial dysfunction and environmental toxicant exposures. Mol Psychiatry. 2012 Apr;17(4):389-401. doi: 10.1038/mp.2011.165. Epub 2011 Dec 6. PMID 22143005
- [Background] Schieve LA, Blumberg SJ, Rice C, Visser SN, Boyle C. The relationship between autism and parenting stress. Pediatrics. 2007 Feb;119 Suppl 1:S114-21. doi: 10.1542/peds.2006-2089Q. PMID 17272578
- [Background] Singh K, Connors SL, Macklin EA, Smith KD, Fahey JW, Talalay P, Zimmerman AW. Sulforaphane treatment of autism spectrum disorder (ASD). Proc Natl Acad Sci U S A. 2014 Oct 28;111(43):15550-5. doi: 10.1073/pnas.1416940111. Epub 2014 Oct 13. PMID 25313065